CLINICAL TRIAL: NCT02702297
Title: Multimodales Monitoring Des Fetalen Inflammationsrisikos Bei frühem Vorzeitigen Blasensprung (PPROM)
Brief Title: Multimodal Monitoring of Fetal Risk of Inflammation in Preterm Premature Rupture of Membranes
Acronym: MuMFI-PPROM
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Jena University Hospital (Other); University of Leipzig (Other); St. Elisabeth Hospital Halle (Unknown)
Responsible Party: Principal Investigator, Gregor Seliger, Dr. med.; chief resident, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: MuMFI-PPROM
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Preterm Premature Rupture of Membranes; Fetal Inflammatory Response Syndrome; Early Onset Neonatal Sepsis; Infection of Amniotic Cavity
Keywords: Preterm premature rupture of the membranes; PPROM; PROM; fetal membranes; premature rupture; neonatal early onset sepsis; amniotic fluid; amniotic infection; fetal inflammatory response syndrome; adverse neonatal outcome; FIRS
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; fetal inflammatory response syndrome; Neonatal Sepsis; Chorioamnionitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: daily multimodal monitoring during pregnancy after PPROM, Analysis of neonatal routine parameters and histologic examination of placenta
  Interventions: Other: single arm

INTERVENTIONS:
Other: single arm — Daily monitoring of vaginal fluid IL6 and fetal ECG. Daily maternal monitoring and delivery according to standard operating procedure. Post partum diagnosis of FIRS or EOS by analysing of fetal cord blood IL6 and clinical signs of sepsis. Diagnosis of histologic amniotic infection by histological analysis.

SUMMARY:
The purpose of this study is to examine whether the value of vaginal fluid cytokine levels as well as computerized fetal ECG analysis are suitable clinical parameters to detect an imminent intra-amniotic inflammation with a high risk of fetal inflammatory response syndrome (FIRS) or a neonatal early onset sepsis (EOS) and whether these parameters can be determined on a daily basis in the clinical monitoring of pregnancies complicated by PPROM.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) is one of the leading causes for preterm birth and adverse neonatal outcome. Between 24 0/7 and 34 0/7 weeks of gestation the prolongation of pregnancy is the recommended course of action to reduce the risks of prematurity in most countries. An intra-amniotic infection resulting in fetal inflammatory response syndrome (FIRS) or early onset neonatal sepsis (EOS) is often associated with high morbidity and mortality.

Standard monitoring includes the maternal response to inflammation (i.e. maternal serum parameters) as well as fetal signs of acute FIRS (i.e. fetal tachycardia, high cytokine level in amniotic fluid obtained by amniocentesis). Changes of fetal ECG-parameters are also a sign of an acute FIRS.

Currently, there is no adequate parameter for the surveillance of a possible ongoing intra-amniotic infection. Other studies have reported a correlation between vaginal fluid interleukine 6 (IL6) collected noninvasively and the risk of FIRS and EOS. Information obtained by computerized fetal ECG analysis might be suitable to detect early signs of fetal infection before the manifestation of FIRS.

With the implementation of a vaginal fluid collector it is possible to detect the vaginal fluid cytokine in clinical everyday routine. With the improvement of fetal ECG monitoring it is possible to record the fetal ECG daily. This study examines the correlation between these new parameters and the onset of fetal infection before the manifestation of a severe systemic fetal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of preterm rupture of the fetal membranes
* Pregnancy between 24 0/7 and 34 0/7 weeks of gestation
* Ability to give informed consent in german or english

Exclusion Criteria:

* Sign of acute amniotic infection syndrome
* independent indication for urgent delivery
* Active labor
* Missing informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with PPROM-complicated pregnancies who referre to one of the participating tertiary referreal care centers.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Odds ratio for severe fetal/early onset neonatal Infection | postpartum one point assessment/ first three days post partum
  combined outcome - rate of: early onset neonatal sepsis, elevated IL6 concentration in cord blood sample, histological signs of funisitis

SECONDARY OUTCOMES:
combined neonatal adverse outcome | 28 days
  rate of severe intraventricular hemorrhage, necrotizing enterocolitis, late onset sepsis, white matter damage within the first 28 days of life
late onset neonatal sepsis | 28 days
  clinical Sepsis after first 72h of life
Severe neonatal cerebral hemorrhage | 28 days
  IVH II+IV°
necrotizing enterocolitis | 28 days
  NEC
umbilical cord blood IL 6 concentration | first day after delivery
  IL-6-concentration in cord blood sample after delivery or in fetal Serum during first hour of life
neonatal early onset sepsis | 3 days
  clinical Sepsis during first 72h of life
histological funisitis | first day after delivery
  redline maternal stage >1, fetal stage >0

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Seliger, Dr. med, Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Michael Bergner, Principal Investigator — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Uwe Schneider, Prof., Principal Investigator — Maternity Clinic; Jena University Hospital; Michael Tchirikov, Prof., Study Chair — Maternity Clinic/Perinatal Treatment Center, Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Frank Bernhard Kraus, PD; PhD, Principal Investigator — Department of Laboratory Medicine; Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Roland Haase, PD, Principal Investigator — Department of Pediatrics; Halle university hospital, Martin-Luther-Universität Halle-Wittenberg; Holger Stepan, Prof., Principal Investigator — Maternity clinic, University of Leipzig
Locations (4):
- Germany (4):
  - Maternity clinic, University of Leipzig, Leipzig, Saxony
  - St. Elisabeth Hospital Halle, Halle, Saxony-Anhalt
  - Maternity Clinic/Perinatal Treatment Center, university hospital, Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Maternity Clinic, Jena University Hospital, Jena, Thuringia